CLINICAL TRIAL: NCT03795285
Title: The Role of Neutrophil CD64 and Soluble Triggering Receptor Expressed on Myeloid Cells 1 in Neonatal Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham I El-mahdy, Principal Investigator, Assiut University
Other Study IDs: Neonatal sepsis
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Neonatal SEPSIS
Keywords: Early onset sepsis; sTREM-1; Neutrophil CD64
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Septic neonates:: fifty neonates with sepsis.
  Interventions: Diagnostic Test: Expression of neutrophil CD64
- Controls:: twenty healthy neonates.
  Interventions: Diagnostic Test: Expression of neutrophil CD64

INTERVENTIONS:
Diagnostic Test: Expression of neutrophil CD64 — Expression of neutrophil CD64 will be measured by Flow cytometry. In addition, sTREM-1 will be measured in the serum by ELISA

SUMMARY:
Neonatal sepsis (NS) is a rather serious but relatively common health problem. Despite recent advances in the treatment of neonatal infection, mortality and comorbidities remain high.

DETAILED DESCRIPTION:
Neonatal sepsis is a major contributor to an estimated 2.6 million annual deaths and accounts for approximately 3 % of all disability-adjusted life years. The consequences of NS can be minimized by early initiation of antibiotic therapy. Due to high NS rates, the vulnerability of the organism in the neonatal period and concerns about consequences (considerable mortality, association with other acute or chronic complications), antibiotic therapy is com¬monly started in clinical practice even though non-spe¬cific clinical signs develop. This is in spite of the fact that antibiotic overuse is linked to major negative outcomes. The reliable and early diagnosis of NS is therefore essential but, unfortunately, rather difficult.

Probably the most widely used "biochemical" marker of NS, C-reactive protein (CRP), is one of the so-called late markers. Its sensitivity is mainly low in the early stages of infection; its reliability increases, particularly with serial measurements. In that case, its negativity practically rules out the presence of NS. It is not completely specific for NS. Procalcitonin (PCT), an intermediate marker, is relatively specific, providing prognostic information as well; it decreases rapidly in response to effective therapy. However, its complex postnatal "physiological" dynamics makes its measurements difficult, particularly in early-onset sepsis.

CD64 is normally expressed in very low concentrations by unstimulated neutrophils. It is considerably upregulated on the trigger of bacterial invasion and has been shown to be involved in the process of phagocytosis and intracellular killing of pathogens. More importantly, neutrophils from preterm infants express CD64 during bacterial infections to the same degree as those from term infants, children, and adults. So in newborns, neutrophil CD64 have been found to be promising markers for diagnosis of early and late infections.

Among several candidate receptors, triggering Receptor Expressed on Myeloid cells 1 (TREM-1) appears to play a relevant role in the modulation of innate immunity, amplifying or attenuating Toll-Like Receptor (TLR)-induced signals. TREM-1 is a receptor of the immunoglobulin superfamily, expressed on human neutrophils and monocytes. In the early phase of infection, the engagements of Pattern Recognition Receptors (PRRs) by microbial components induce up-regulation of TREM-1. After recognition of a still unknown ligand, TREM-1 associates with a signal transduction molecule called DAP12, triggering the sustained release of pro-inflammatory cytokines (TNF-alpha and IL-1b) and chemokines (IL-8 and monocyte chemotactic protein), which may result in prolonged survival of neutrophils and monocytes at the inflammatory site.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis was defined as a positive blood culture in infants with clinical and laboratory findings of infection. Manifestations of sepsis include poor suckling, sleepiness, respiratory distress, apnea, poor perfusion, cyanosis, bradycardia, fever or hypothermia, feeding intolerance, and neurological signs (as seizures). Routine sepsis evaluations included complete blood count, C-reactive protein, and blood culture.

Exclusion Criteria:

* malformations
* prematurity
* Apgar score less than seven
* on antibiotics treatment before the start of the study

Ages: 1 Day to 50 Days | Sex: All
Age Groups: Child
Study Population: Neonatal sepsis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-02-20 (Estimated); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-09-30 (Estimated)

PRIMARY OUTCOMES:
The mean difference of neutrophil CD64 expression and sTREM-1 before and after treatment | 72 hours
  better understanding of neutrophil CD64 role as an essential player in pathogenesis of neonatal sepsis and the role of and sTREM-1 in pathogenesis of neonatal sepsis

REFERENCES:
- [Background] Halek J, Novak M, Medkova A, Furst T, Juranova J. The role of nCD64 in the diagnosis of neonatal sepsis in preterm newborns. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2018 Jun 21. doi: 10.5507/bp.2018.033. Online ahead of print. PMID 29955185
- [Background] Wright JK, Hayford K, Tran V, Al Kibria GM, Baqui A, Manajjir A, Mahmud A, Begum N, Siddiquee M, Kain KC, Farzin A. Biomarkers of endothelial dysfunction predict sepsis mortality in young infants: a matched case-control study. BMC Pediatr. 2018 Mar 23;18(1):118. doi: 10.1186/s12887-018-1087-x. PMID 29571293
- [Background] Ford JW, McVicar DW. TREM and TREM-like receptors in inflammation and disease. Curr Opin Immunol. 2009 Feb;21(1):38-46. doi: 10.1016/j.coi.2009.01.009. Epub 2009 Feb 21. PMID 19230638
- [Background] Groselj-Grenc M, Ihan A, Derganc M. Neutrophil and monocyte CD64 and CD163 expression in critically ill neonates and children with sepsis: comparison of fluorescence intensities and calculated indexes. Mediators Inflamm. 2008;2008:202646. doi: 10.1155/2008/202646. PMID 18604302